CLINICAL TRIAL: NCT04712318
Title: Succesful Treatment of Residual Refraction Errors (Myopic and Hyperopic) 6 Months After Trifocal IOL Implantation With Relex-Smile
Brief Title: Treatment of Residual Refraction Errors 6 Months After Trifocal IOL Implantation With Relex-Smile
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHospitalPristina
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pseudophakia; Myopia; Hyperopia
MeSH Terms: conditions — Pseudophakia; Myopia; Hyperopia

STUDY DESIGN:
Intervention Model Description: Myopic group 100 eyes hyperopic group 30 eyes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReLex Smile surgery (Other): The aim of this study is to investigate the effect of Relex Smile surgery to correct the residual refractive errors (myopic and hyperopic) 6 months after Trifocal IOL Implantation.
  At myopic residual refraction (min -0.75 D) (100eyes) 6 months after Trifocal IOL Implantation we used Relex-Smile surgery for treatment.
  Interventions: Procedure: Relex Smile
- ReLex Smile surgery-fresh corneal lenticule implantation (Other): At hyperopic residual refraction 30 eyes 6 months after Trifocal IOL Implantation we used fresh corneal myopic lenticule implantation as allogenic implant that will be taken from myopic patients to implant on pseudophakic patients with residual hypermetropic refraction using VisuMax Femtosecond Laser-Smile module surgery with primary objective to assess(increase) visual acuity.
  Interventions: Procedure: Relex smile with fresh corneal lenticule implantation

INTERVENTIONS:
Procedure: Relex Smile — Procedure/Surgery: Relex Smile The residual myopic refraction on Pseudophakic patients after 6 months using Relex-Smile surgery by VisuMax femtosecond laser. The residual refractive power was min -0.75D.The optical zone (lenticule diameter) and cap diameter were 6.5 and 7.5 mm respectively. After dissection of both anterior and posterior planes, the lenticule was extracted through 120 degree superior 3.5 mm incision and marked with a sterile marker(ViscotMedster).
  Arms: ReLex Smile surgery
Procedure: Relex smile with fresh corneal lenticule implantation — VisuMax femtosecond laser performed flap-cut procedure with an energy cut index of 30 nJ (150nJ), spot and track spacing surface cut of 4.5 μm, side cut 2.0 μm were used to create an intrastromal pocket into the patient's cornea to receive the donor lenticule.
  The stromal pocket diameter was set 7.6 to 8.0 mm (1 mm larger than the optical zone of the donor lenticule) and cap thickness was set to 130 μm from corneal surface and a 4 mm superior incision. Hinge position flap was set at 90°, angle 50° and width 4 mm, side cut angle 90°. The pocket was dissected using a blunt spatula washed with normal saline. The lenticule was held with lenticule forceps and gently inserted into the pocket through the 4 mm superior incision.
  In pseudophakic patients with hyperopic astigmatism residual refraction, corneal topography-guided intrastromal fresh lenticular implantation should be performed according to the low K values.
  Arms: ReLex Smile surgery-fresh corneal lenticule implantation

SUMMARY:
Successful treatment of residual refraction 6 months after IOL Implantation with Relex-Smile.

DETAILED DESCRIPTION:
Residual refractive errors(myopia 50% and hyperopia 30%) are the main problems at patients after IOL Implantation.

The residual refraction (myopic and hyperopic) after IOL Implantation is difficult to treat surgically. In addition, there are not many suitable options to offer such patients presenting with this condition.

Two current common surgeries to treat residual hyperopic refraction are refractive lens exchange (RLE) and excimer laser ablation (LASIK or PRK).

Laser procedures: Photorefractive keratectomy (PRK); Laser assisted in situ keratomileusis (LASIK); Risks of LASIK include abnormalities of the corneal flap, epithelial ingrowth, corneal ectasia, refractive surprises, irregular astigmatism, decentration, visual aberrations, a loss of BCVA, infectious keratitis, symptoms, and diffuse lamellar keratitis.

Refractive lens exchange (RLE); The risks of RLE are similar to those of cataract surgery and include endophthalmitis, a loss of accommodation, vitreous loss with posterior capsular rupture, and retinal detachment.

The aim of our study is to investigate the effect of Relex-Smile to treat the residual refraction errors (myopia and hypermetropia) 6 months after IOL Implantation.

Before SMILE, Yag-Laser capsulotomy should be performed on all patients, regardless of posterior capsule ossification, in pseudophakic patients with residual refraction. When the YAG Laser is applied after the SMILE ,there will be a diopter change. In pseudophakic patients with hyperopic astigmatism and residual refraction ,corneal topography-guided intrastromal fresh lenticular implantation should be performed and the lenticule was placed according to the low K value.

At myopic residual refraction(-0.75D till -5.50D) after IOL Implantation The method used at the EYE Hospital Pristina by ReLex-SMILE is safe and effective method, since there is no flap and this prevents invasive damage to the anterior surface of the cornea contrary to the LASIK where flap is present posing risk for epithelial ingrowth.

At hyperopic residual refraction this study is to investigate the effect of fresh myopic corneal lenticule implantation as allogenic implant(-1.50D) that will be taken from myopic patients to implant on Pseudophakic patients with residual hypermetropia refraction (+1.0D) using VisuMax Femtosecond laser - Smile module surgery

ELIGIBILITY:
Inclusion Criteria:

* residual hypermetropic, myopic refraction on pseudophakic patients
* low visual acuity

Exclusion Criteria:

* active anterior segment pathologic features,
* previous corneal or anterior segment surgery,
* glaucoma,
* retinal detachment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Increase of visual acuity | 6 months
  Increase of visual acuity by reducing residual refractive errors (myopia, hyperopia) using ReLex Smile after Trifocal IOL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo